CLINICAL TRIAL: NCT04200573
Title: A Phase 1, Open-Label, Single Dose Study to Evaluate the Pharmacokinetics of Ampreloxetine Following a Single-dose in Subjects With Mild, Moderate, and Severe Hepatic Impairment and in Matching Healthy Subjects
Brief Title: Effect of Hepatic Impairment on the Pharmacokinetics of a Single Dose of TD-9855
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Theravance Biopharma (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 0179
Record Dates: First submitted 2019-12-13; First posted 2019-12-16 (Actual); Last update posted 2021-09-08 (Actual); Status verified 2021-09

CONDITIONS: Symptomatic Neurogenic Orthostatic Hypertension; nOH
Keywords: Symptomatic neurogenic orthostatic hypertension; hepatic impairment
MeSH Terms: interventions — ampreloxetine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Normal Hepatic Function (Experimental): Ampreloxetine Dose A single dose administration to subjects with normal hepatic function
  Interventions: Drug: Ampreloxetine
- Mild Hepatic Function (Experimental): Ampreloxetine Dose A single dose administration to subjects with mild hepatic impairment
  Interventions: Drug: Ampreloxetine
- Moderate Hepatic Function (Experimental): Ampreloxetine Dose A single dose administration to subjects with moderate hepatic impairment
  Interventions: Drug: Ampreloxetine
- Severe Hepatic Function (Experimental): Ampreloxetine Dose A single dose administration to subjects with severe hepatic impairment
  Interventions: Drug: Ampreloxetine

INTERVENTIONS:
Drug: Ampreloxetine — The study drug will be administered orally as a single Dose A tablet
  Other Names: TD-9855

SUMMARY:
An open-label study to characterize the effects of mild, moderate, and severe Hepatic Impairment (HI) on the pharmacokinetics (PK) of ampreloxetine following a single oral dose in comparison with healthy volunteers with normal hepatic function.

DETAILED DESCRIPTION:
This is a multicenter, non-randomized, open label, parallel group, single dose, 2-part study being conducted in adult subjects with mild, moderate, or severe HI (Child-Pugh Class A, B, and C), and in matching healthy subjects. The healthy matching group will be comparable to the corresponding hepatic impairment groups by matching subjects by weight (±20% of group mean), age (±10 years of group mean), and sex (equal ratios across groups).

The study will be conducted in two sequential parts:

In Part A, following a 28-day screening period, 6 subjects each with mild or moderate HI and 6 matching healthy subjects who meet eligibility criteria will be enrolled and administered a single Dose A (Day 1).

In Part B, following a 28-day screening period, 6 subjects with severe hepatic impairment will receive a single Dose A (Day 1). Furthermore, the Sponsor may choose to enroll up to 6 additional healthy subjects in Part B to ensure matching of subjects across all groups for weight, age, and sex is maintained.

ELIGIBILITY:
Inclusion Criteria:

All Subjects:

* has a body mass index (BMI) of 19 to 40 kg/m2, inclusive, and weight of at least 55 kg.
* clinical labs within normal ranges
* creatinine clearance of >70 mL/min
* women must be non-pregnant and non-lactating, male and females must agree to highly effective methods of contraception
* additional criteria apply

Subjects with Impaired Hepatic Function additional criteria:

* Subject has mild (Child-Pugh Class A [5 to 6 points]), moderate (Child-Pugh Class B [7 to 9 points]), or severe (Child-Pugh Class C [10-15 points]) liver disease
* has stable hepatic impairment defined as no clinically significant change in disease status within the last 30 days
* must be on a stable dose of medication and/or treatment regimen at least 30 days before dosing
* Additional inclusion criteria apply

Exclusion Criteria:

Subjects with normal hepatic function:

* history of reactions or hypersensitivity to ampreloxetine or known intolerance to other norepinephrine reuptake inhibitors (NRI) or serotonin norepinephrine reuptake inhibitors (SNRI).
* personal or family history of congenital long QT syndrome
* history of untreated closed angle glaucoma
* history of orthostatic hypotension or orthostatic tachycardia or a history of dizziness, lightheadedness or fainting, or a feeling of blacking out upon standing
* has used nephrotoxic or hepatotoxic medications 30 days before Day-2
* routinely uses more than 2 grams of acetaminophen daily
* has used tobacco-containing products (e.g., cigarettes, cigars, chewing tobacco, snuff, e cigarettes, vaporizers) within 3 months before Screening or has a positive cotinine result at Screening or Day -2
* used any CYP1A2 inhibitor or inducer within 7 days or 5 half lives, whichever is longer, prior to ampreloxetine dosing or requires concomitant use
* has used monoamine oxidase inhibitors (MAO-I) within 7 days or 5 half lives, whichever is longer, prior to ampreloxetine dosing or requires concomitant use
* additional exclusion criteria apply

Subjects with impaired hepatic function additional criteria:

* has severe ascites that could potentially interfere with respiratory function
* current severe hepatic encephalopathy
* history of liver transplantation, hepatocellular carcinoma, or acute liver disease
* has biliary liver cirrhosis
* has uncontrolled hypertension (SBP >180 mm Hg and DBP (Diastolic blood pressure) >110 mm Hg)
* has an abnormal ECG at Screening or Day -2, including QTcF (Fridericia's corrected QT Interval) >470 msec
* additional exclusion criteria apply

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 31 (Actual)
Dates: Start 2020-01-13 (Actual); Primary Completion 2021-08-19 (Actual); Study Completion 2021-08-19 (Actual)

PRIMARY OUTCOMES:
Plasma AUC0-t | Plasma AUC0-t will be measured Day 1 to Day 15
  Estimation of Area under the concentration-time curve, from time zero to the last measured time point
Plasma AUC0-inf | Plasma AUC0-inf will be measured from Day 1 to Day 15
  Estimation of AUC from time zero extrapolated to infinity
Plasma Cmax | up to Day 21
  Estimation of maximum observed plasma concentration

SECONDARY OUTCOMES:
Number of subjects with clinically significant vital sign abnormalities | up to Day 21
  Clinically significant abnormalities in vital signs will be listed and described
Number of subjects with change in C-SSRS scores | up to Day 21
  Changes in Columbia suicide severity rating scale (C-SSRS) scores will be listed and described

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Theravance Biopharma
Locations (2):
- United States (2):
  - Theravance Biopharma Investigational Site, Miami, Florida
  - Theravance Biopharma Investigational Site, Orlando, Florida

IPD SHARING:
Plan to Share IPD: No
Theravance Biopharma, Inc. will not be sharing individual de-identified participant data or other relevant study documents.

REFERENCES:
- [Derived] Kanodia J, Giovinazzo H, Yates W, Bourdet DL, McRae MP, Helmke SM, Everson GT. Hepatic Dysfunction Quantified by HepQuant DuO Outperforms Child-Pugh Classification in Predicting the Pharmacokinetics of Ampreloxetine. Clin Pharmacol Ther. 2024 Jul;116(1):186-193. doi: 10.1002/cpt.3265. Epub 2024 Apr 23. PMID 38654484